CLINICAL TRIAL: NCT05341271
Title: The Effect of Digital Reminiscence Therapy on People With Mild and Moderate Dementia: A Randomized Controlled Trial.
Brief Title: The Effect of Digital Reminiscence Therapy on People With Mild and Moderate Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJU-IRB C110100
Record Dates: First submitted 2022-03-08; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Dementia
Keywords: dementia; digital technology; reminiscence group; neuropsychiatric symptoms; depression, life meaning; caregiver burden
MeSH Terms: conditions — Dementia; Depression; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital reminiscence group (DRG) (Other): Experiment group A accepted the planned digital nostalgic group activities using the official account platform of line as a medium, one class per week, 45-50 minutes each time, lasting 8 times.
  Interventions: Other: Experimental: digital reminiscence group (DRG)
- general reminiscence group (GRG) (Other): Experiment group B participated in a general traditional nostalgic group, using actual nostalgic objects or utensils to carry out nostalgic activities, one class per week, 45-50 minutes each time, lasting 8 times
  Interventions: Other: Experimental: general reminiscence group (GRG)

INTERVENTIONS:
Other: Experimental: digital reminiscence group (DRG) — Experiment group A accepted the digital reminiscence group planned by the official account platform of line as the medium, the theme and content, it is planned to consider the development of the life cycle, and the experience of the thematic review will induce the motivation of the participants, since childhood life, study The design of eight unit themes such as stage, work and emotional family and festival life, and special life events; at the same time, it can adapt to the psychological adaptation behavior of the participants, review their life development stages according to the life development process, and pay attention to the interpersonal interaction carried out by the current group Negative emotional or symptomatic behavior with dialogue, and directing and dealing with life experiences
  Arms: digital reminiscence group (DRG)
Other: Experimental: general reminiscence group (GRG) — Experiment group B participated in general reminiscence group (GRG)
  , using actual nostalgic objects or utensils to carry out activities. The theme and content are intended to be considered in the context of life cycle development, and the experience of thematic retrospectives induces the motivation of participants, since childhood. The design of eight unit themes, including the stage of study, work and emotional family and festival life, and special events in life; at the same time, it can adapt to the psychological adaptation behavior of the participants, review their life development stages according to the life development process, and pay attention to the current group activities. Interpersonal interaction and dialogue, and negative emotional or symptomatic behaviors that guide and process life experiences
  Arms: general reminiscence group (GRG)

SUMMARY:
In the post-epidemic era, it is necessary to develop support programs for families with dementia in empirical care. The reminiscence therapy was adopted by patients with mild and moderate dementia those intervention have had good memory stimulation and emotional support effects in the previous studies. However, the application of digital reminiscence therapy that cross spatial and geographic constraints, but related research still has limitations on the knowledge of this topic.

To use the official Line @ account as a media platform to develop a digital reminiscence group program (DRG), and to investigate the effects of mobile-application-based DRG on the psychoneurological symptoms, depression, life meaning and burden of family caregiver in people with mild and moderate dementia (PMMD).

DETAILED DESCRIPTION:
In the post-epidemic era, it is necessary to develop support programs for families with dementia in empirical care. The reminiscence therapy was adopted by patients with mild and moderate dementia those intervention have had good memory stimulation and emotional support effects in the previous studies. However, the application of digital reminiscence therapy that cross spatial and geographic constraints, but related research still has limitations on the knowledge of this topic.

To use the official Line @ account as a media platform to develop a digital reminiscence group program (DRG), and to investigate the effects of mobile-application-based DRG on the psychoneurological symptoms, depression, life meaning and burden of family caregiver in people with mild and moderate dementia (PMMD).

This will be the first digital reminiscence group constructed specifically for family's people with mild and moderate dementia in our country. The investigators expected to have a positive effect. It can be used as a reference for the development of empirical care programs for family caregivers with PMMD in the community.

ELIGIBILITY:
Inclusion Criteria:

* The conditions for accepting cases for families with dementia are as follows:

  1. Family caregivers must meet the following conditions:

     ①Age 20 years old or above

     ②Have experience in caring for the dementia case in the past year, and live together
     * Have a smart phone and have experience in using line APP
  2. Dementia patients must meet the following conditions:

     * Those who currently live at home and regularly go to the Rizhao Center to participate in activities ②Patients with dementia (Alzheimer's disease) diagnosed by a physician with DSM 5 or in line with NINCDS/ADRDA, their CDR score is 1~2 points ③ Those who have a clear consciousness, can express in Chinese and Taiwanese, or communicate with others in words without hindrance ④ Those who have normal vision and hearing, and can operate digital mobile phones or tablets

Exclusion Criteria:

* The exclusion criteria for families with dementia are:

  1. The exclusion conditions for family caregivers are:

     * A history of mental illness diagnosed by a psychiatrist, such as major depression ② Those who are not of their own nationality.
  2. The exclusion conditions for patients with dementia are:

     * Confusion or delirium ② Dementia cases who will be referred to long-term care institutions or nursing homes within one month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination; MMSE | Pre-intervention(T0)
  The content of the test includes orientation, immediate memory, recent memory, concentration or attention, etc. The full score is 30 points. It is currently used in clinical and research, and is often used for cognitive evaluation of the elderly, and is widely used.
Neuropsychiatric Inventory, NPI | Pre-intervention(T0)
  The content of the scale is to ask primary caregivers about new behaviors or changes in behavior since the onset of the patient, whether in the past four weeks or within a specified period of time. NPI includes 12 psycho-behavioral symptom items. The scoring method first uses screening questions to determine whether there is a change in behavior, then in-depth understanding of the changed behavior, and finally determines the frequency, severity and caregiver distress of the behavior according to each behavior degree. In terms of reliability and validity of the scale, the Cronbach's alpha for Chinese was 0.76, and the test-retest reliabilities of severity frequency and caregiver stress in the scale were 0.82, 0.85 and 0.79 respectively. It also has good reliability and validity (Fuh, Liu, Mega, Wang, & Cummings, 2001), and the assessment source of this scale is mainly asking the family caregivers of the patients.
Cornell Scale for Depression in Dementia; CSDD | Pre-intervention(T0)
  For patients with dementia who cannot communicate properly with others through oral expressions, making it difficult to identify their depressive symptoms, the application of this observation scale can effectively and appropriately detect depression in the elderly with cognitive impairment. The Kappa value of the two-week rater-ask agreement reliability (inter-rater agreement) was .43, indicating that all items were significantly stable; and the Cronbach's alpha of the internal consistency reliability was .84, this scale The source of the assessment was primarily asking the patient's family caregiver.
Purpose in Life Test: | Pre-intervention(T0)
  This scale is used to assess the extent to which the elderly perceive the meaning and purpose of their life. There are 9 questions in two aspects (personal value and success of children and grandchildren), which are answered on a four-point scale. Among them, questions 5 and 6 are reverse questions. The total score ranges from 9 to 36 points. The higher the total score, the more positive and meaningful the subject feels about life. This scale has content validity completed by experts and scholars, and the internal consistency Cronbach α value of the scale is .75. After factor analysis, the explained variation of the two factors of shaping can reach 54.4%, indicating that this scale has good performance. reliability and validity.
Mini-Mental State Examination; MMSE | two momths after intervention(T1)
  The content of the test includes orientation, immediate memory, recent memory, concentration or attention, etc. The full score is 30 points. It is currently used in clinical and research, and is often used for cognitive evaluation of the elderly, and is widely used.
Neuropsychiatric Inventory, NPI | two momths after intervention(T1)
  The content of the scale is to ask primary caregivers about new behaviors or changes in behavior since the onset of the patient, whether in the past four weeks or within a specified period of time. NPI includes 12 psycho-behavioral symptom items. The scoring method first uses screening questions to determine whether there is a change in behavior, then in-depth understanding of the changed behavior, and finally determines the frequency, severity and caregiver distress of the behavior according to each behavior degree. In terms of reliability and validity of the scale, the Cronbach's alpha for Chinese was 0.76, and the test-retest reliabilities of severity frequency and caregiver stress in the scale were 0.82, 0.85 and 0.79 respectively. It also has good reliability and validity (Fuh, Liu, Mega, Wang, & Cummings, 2001), and the assessment source of this scale is mainly asking the family caregivers of the patients.
Cornell Scale for Depression in Dementia; CSDD | two momths after intervention(T1)
  For patients with dementia who cannot communicate properly with others through oral expressions, making it difficult to identify their depressive symptoms, the application of this observation scale can effectively and appropriately detect depression in the elderly with cognitive impairment. The Kappa value of the two-week rater-ask agreement reliability (inter-rater agreement) was .43, indicating that all items were significantly stable; and the Cronbach's alpha of the internal consistency reliability was .84, this scale The source of the assessment was primarily asking the patient's family caregiver.
Purpose in Life Test: | two momths after intervention(T1)
  This scale is used to assess the extent to which the elderly perceive the meaning and purpose of their life. There are 9 questions in two aspects (personal value and success of children and grandchildren), which are answered on a four-point scale. Among them, questions 5 and 6 are reverse questions. The total score ranges from 9 to 36 points. The higher the total score, the more positive and meaningful the subject feels about life. This scale has content validity completed by experts and scholars, and the internal consistency Cronbach α value of the scale is .75. After factor analysis, the explained variation of the two factors of shaping can reach 54.4%, indicating that this scale has good performance. reliability and validity.
Mini-Mental State Examination; MMSE | One month after the end of the intervention (T2)
  The content of the test includes orientation, immediate memory, recent memory, concentration or attention, etc. The full score is 30 points. It is currently used in clinical and research, and is often used for cognitive evaluation of the elderly, and is widely used.
Neuropsychiatric Inventory, NPI | One month after the end of the intervention (T2)
  The content of the scale is to ask primary caregivers about new behaviors or changes in behavior since the onset of the patient, whether in the past four weeks or within a specified period of time. NPI includes 12 psycho-behavioral symptom items. The scoring method first uses screening questions to determine whether there is a change in behavior, then in-depth understanding of the changed behavior, and finally determines the frequency, severity and caregiver distress of the behavior according to each behavior degree. In terms of reliability and validity of the scale, the Cronbach's alpha for Chinese was 0.76, and the test-retest reliabilities of severity frequency and caregiver stress in the scale were 0.82, 0.85 and 0.79 respectively. It also has good reliability and validity (Fuh, Liu, Mega, Wang, & Cummings, 2001), and the assessment source of this scale is mainly asking the family caregivers of the patients.
Cornell Scale for Depression in Dementia; CSDD | One month after the end of the intervention (T2)
  For patients with dementia who cannot communicate properly with others through oral expressions, making it difficult to identify their depressive symptoms, the application of this observation scale can effectively and appropriately detect depression in the elderly with cognitive impairment. The Kappa value of the two-week rater-ask agreement reliability (inter-rater agreement) was .43, indicating that all items were significantly stable; and the Cronbach's alpha of the internal consistency reliability was .84, this scale The source of the assessment was primarily asking the patient's family caregiver.
Purpose in Life Test: | One month after the end of the intervention (T2)
  This scale is used to assess the extent to which the elderly perceive the meaning and purpose of their life. There are 9 questions in two aspects (personal value and success of children and grandchildren), which are answered on a four-point scale. Among them, questions 5 and 6 are reverse questions. The total score ranges from 9 to 36 points. The higher the total score, the more positive and meaningful the subject feels about life. This scale has content validity completed by experts and scholars, and the internal consistency Cronbach α value of the scale is .75. After factor analysis, the explained variation of the two factors of shaping can reach 54.4%, indicating that this scale has good performance. reliability and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Result] Bejan A, Gundogdu R, Butz K, Muller N, Kunze C, Konig P. Using multimedia information and communication technology (ICT) to provide added value to reminiscence therapy for people with dementia : Lessons learned from three field studies. Z Gerontol Geriatr. 2018 Jan;51(1):9-15. doi: 10.1007/s00391-017-1347-7. Epub 2017 Dec 7. PMID 29218401
- [Result] BUTLER RN. The life review: an interpretation of reminiscence in the aged. Psychiatry. 1963 Feb;26:65-76. doi: 10.1080/00332747.1963.11023339. No abstract available. PMID 14017386
- [Result] Davison TE, Nayer K, Coxon S, de Bono A, Eppingstall B, Jeon YH, van der Ploeg ES, O'Connor DW. A personalized multimedia device to treat agitated behavior and improve mood in people with dementia: A pilot study. Geriatr Nurs. 2016 Jan-Feb;37(1):25-9. doi: 10.1016/j.gerinurse.2015.08.013. Epub 2015 Sep 26. PMID 26412509
- [Result] Etters L, Goodall D, Harrison BE. Caregiver burden among dementia patient caregivers: a review of the literature. J Am Acad Nurse Pract. 2008 Aug;20(8):423-8. doi: 10.1111/j.1745-7599.2008.00342.x. PMID 18786017
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Fuh JL, Liu CK, Mega MS, Wang SJ, Cummings JL. Behavioral disorders and caregivers' reaction in Taiwanese patients with Alzheimer's disease. Int Psychogeriatr. 2001 Mar;13(1):121-8. doi: 10.1017/s1041610201007517. PMID 11352329
- [Result] Huang HC, Chen YT, Chen PY, Huey-Lan Hu S, Liu F, Kuo YL, Chiu HY. Reminiscence Therapy Improves Cognitive Functions and Reduces Depressive Symptoms in Elderly People With Dementia: A Meta-Analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2015 Dec;16(12):1087-94. doi: 10.1016/j.jamda.2015.07.010. Epub 2015 Sep 1. PMID 26341034
- [Result] Joddrell P, Astell AJ. Studies Involving People With Dementia and Touchscreen Technology: A Literature Review. JMIR Rehabil Assist Technol. 2016 Nov 4;3(2):e10. doi: 10.2196/rehab.5788. PMID 28582254
- [Result] Jones C, Sung B, Moyle W. Engagement of a Person with Dementia Scale: Establishing content validity and psychometric properties. J Adv Nurs. 2018 May 17. doi: 10.1111/jan.13717. Online ahead of print. PMID 29772602
- [Result] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Result] Laver K, Cumming RG, Dyer SM, Agar MR, Anstey KJ, Beattie E, Brodaty H, Broe T, Clemson L, Crotty M, Dietz M, Draper BM, Flicker L, Friel M, Heuzenroeder LM, Koch S, Kurrle S, Nay R, Pond CD, Thompson J, Santalucia Y, Whitehead C, Yates MW. Clinical practice guidelines for dementia in Australia. Med J Aust. 2016 Mar 21;204(5):191-3. doi: 10.5694/mja15.01339. PMID 26985848
- [Result] Lazar A, Thompson H, Demiris G. A systematic review of the use of technology for reminiscence therapy. Health Educ Behav. 2014 Oct;41(1 Suppl):51S-61S. doi: 10.1177/1090198114537067. PMID 25274711
- [Result] Liu Y, Yan LM, Wan L, Xiang TX, Le A, Liu JM, Peiris M, Poon LLM, Zhang W. Viral dynamics in mild and severe cases of COVID-19. Lancet Infect Dis. 2020 Jun;20(6):656-657. doi: 10.1016/S1473-3099(20)30232-2. Epub 2020 Mar 19. No abstract available. PMID 32199493
- [Result] Lorenz K, Freddolino PP, Comas-Herrera A, Knapp M, Damant J. Technology-based tools and services for people with dementia and carers: Mapping technology onto the dementia care pathway. Dementia (London). 2019 Feb;18(2):725-741. doi: 10.1177/1471301217691617. Epub 2017 Feb 8. PMID 28178858
- [Result] Marshall F, Gordon A, Gladman JRF, Bishop S. Care homes, their communities, and resilience in the face of the COVID-19 pandemic: interim findings from a qualitative study. BMC Geriatr. 2021 Feb 5;21(1):102. doi: 10.1186/s12877-021-02053-9. PMID 33546612
- [Result] Martinsson L, Strang P, Bergstrom J, Lundstrom S. Dying from COVID-19 in nursing homes-sex differences in symptom occurrence. BMC Geriatr. 2021 May 6;21(1):294. doi: 10.1186/s12877-021-02228-4. PMID 33957890
- [Result] McCauley CO, Bond RB, Ryan A, Mulvenna MD, Laird L, Gibson A, Bunting B, Ferry F, Curran K. Evaluating User Engagement with a Reminiscence App Using Cross-Comparative Analysis of User Event Logs and Qualitative Data. Cyberpsychol Behav Soc Netw. 2019 Aug;22(8):543-551. doi: 10.1089/cyber.2019.0076. PMID 31403855
- [Result] Moon S, Park K. The effect of digital reminiscence therapy on people with dementia: a pilot randomized controlled trial. BMC Geriatr. 2020 May 6;20(1):166. doi: 10.1186/s12877-020-01563-2. PMID 32375661
- [Result] Neal I, du Toit SHJ, Lovarini M. The use of technology to promote meaningful engagement for adults with dementia in residential aged care: a scoping review. Int Psychogeriatr. 2020 Aug;32(8):913-935. doi: 10.1017/S1041610219001388. Epub 2019 Sep 24. PMID 31547900
- [Result] GBD 2016 Dementia Collaborators. Global, regional, and national burden of Alzheimer's disease and other dementias, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Jan;18(1):88-106. doi: 10.1016/S1474-4422(18)30403-4. Epub 2018 Nov 26. PMID 30497964
- [Result] Park K, Lee S, Yang J, Song T, Hong GS. A systematic review and meta-analysis on the effect of reminiscence therapy for people with dementia. Int Psychogeriatr. 2019 Nov;31(11):1581-1597. doi: 10.1017/S1041610218002168. Epub 2019 Feb 4. PMID 30712519
- [Result] Penning MJ, Wu Z. Caregiver Stress and Mental Health: Impact of Caregiving Relationship and Gender. Gerontologist. 2016 Dec;56(6):1102-1113. doi: 10.1093/geront/gnv038. Epub 2015 Apr 17. PMID 26035875
- [Result] Robinson L, Clare L, Evans K. Making sense of dementia and adjusting to loss: psychological reactions to a diagnosis of dementia in couples. Aging Ment Health. 2005 Jul;9(4):337-47. doi: 10.1080/13607860500114555. PMID 16019290
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Result] Stinson CK. Structured group reminiscence: an intervention for older adults. J Contin Educ Nurs. 2009 Nov;40(11):521-8. doi: 10.3928/00220124-20091023-10. PMID 19904866
- [Result] Subramaniam P, Woods B. Digital life storybooks for people with dementia living in care homes: an evaluation. Clin Interv Aging. 2016 Sep 16;11:1263-1276. doi: 10.2147/CIA.S111097. eCollection 2016. PMID 27698556
- [Result] Tuijt R, Frost R, Wilcock J, Robinson L, Manthorpe J, Rait G, Walters K. Life under lockdown and social restrictions - the experiences of people living with dementia and their carers during the COVID-19 pandemic in England. BMC Geriatr. 2021 May 10;21(1):301. doi: 10.1186/s12877-021-02257-z. PMID 33971847
- [Result] Wang JJ. Group reminiscence therapy for cognitive and affective function of demented elderly in Taiwan. Int J Geriatr Psychiatry. 2007 Dec;22(12):1235-40. doi: 10.1002/gps.1821. PMID 17503545
- [Result] Whitehead BR, Torossian E. Older Adults' Experience of the COVID-19 Pandemic: A Mixed-Methods Analysis of Stresses and Joys. Gerontologist. 2021 Jan 21;61(1):36-47. doi: 10.1093/geront/gnaa126. PMID 32886764
- [Result] Woods B, O'Philbin L, Farrell EM, Spector AE, Orrell M. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2018 Mar 1;3(3):CD001120. doi: 10.1002/14651858.CD001120.pub3. PMID 29493789
- [Result] Woods RT, Bruce E, Edwards RT, Elvish R, Hoare Z, Hounsome B, Keady J, Moniz-Cook ED, Orgeta V, Orrell M, Rees J, Russell IT. REMCARE: reminiscence groups for people with dementia and their family caregivers - effectiveness and cost-effectiveness pragmatic multicentre randomised trial. Health Technol Assess. 2012;16(48):v-xv, 1-116. doi: 10.3310/hta16480. PMID 23211271
- [Result] Yeung DY, Chung EKH, Lam AHK, Ho AKK. Effects of subjective successful aging on emotional and coping responses to the COVID-19 pandemic. BMC Geriatr. 2021 Feb 17;21(1):128. doi: 10.1186/s12877-021-02076-2. PMID 33596829
- [Result] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Result] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- See also: World Health Organization (2021). Dementia. — http://www.who.int/news-room/fact-sheets/detail/dementia